CLINICAL TRIAL: NCT03248349
Title: Population Pharmacokinetics of Antibiotics in Critically Ill Children
Brief Title: Population Pharmacokinetics of Antibiotics in Critically Ill Children (POPSICLE)
Acronym: POPSICLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-3085
Record Dates: First submitted 2017-08-02; First posted 2017-08-14 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2019-09

CONDITIONS: Critical Illness; Infectious Disease; Children
Keywords: Critically ill children; Pharmacokinetics; Anti-Bacterial agents
MeSH Terms: conditions — Critical Illness; Communicable Diseases | interventions — Pharmacokinetics; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood plasma for antibiotic concentrations during admission (max. 14 days)
  * Whole blood sample for future DNA-analysis
  * Urine samples during admission (max. 14 days)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 1: Pharmacokinetics
  Interventions: Drug: Pharmacokinetics

INTERVENTIONS:
Drug: Pharmacokinetics — * Blood samples are drawn for pharmacokinetic properties of antibiotics during routine care treatment
  * Blood samples for relevant covariates of drug disposition (kidney function, liver enzymes, C-reactive protein (CRP), albumin)
  * Whole blood is stored for DNA analysis
  * Urine is drawn from catheter for more detailed estimation of glomerular filtration rate and drug metabolite analysis
  Other Names: Antibiotics

SUMMARY:
Infections are common on the Intensive Care for both adult and pediatric patients. Adequately dosing antibiotic treatment is of vital importance but both under- and overdosing is frequent due to pathophysiological changes during critical illness. Moreover, the interplay of age and critical illness is even more understudied.

To optimize antibiotic dosing and outcome of infectious disease, personalized dosing guidelines in critically ill patients are highly needed. In this prospective observational population pharmacokinetic study we will evaluate if target attainment for antibiotics is reached in critically ill children with current dosing guidelines. Using these data, individualized dosing guidelines will be developed.

DETAILED DESCRIPTION:
Approximately one third of all critically ill children develop infectious disease related complications. Mortality due to infections can be as high as 30-45%. In up to 41% of adult critically ill patients antimicrobial dosing recommendations are inadequate, as acute kidney injury, augmented renal clearance, inflammatory response and hypoalbuminaemia all contribute to variation in drug concentrations. This is an important reason for antibiotic treatment failure and emergence of resistance.

Data from adults cannot be directly extrapolated to children, due to developmental changes in the processes involved in drug disposition. Moreover, the interplay of age and critical illness is even more understudied. Hence, to optimize antibiotic dosing and outcome of infectious disease, personalized dosing guidelines in critically ill patients are highly needed.

In this prospective observational population pharmacokinetic study we will evaluate if target attainment for antibiotics is reached in critically ill children with current dosing guidelines. Using these data, individualized dosing guidelines will be developed.

Objectives:

To determine the population pharmacokinetics of antibiotics in critically ill pediatric patients to develop individualized dosing guidelines for antibiotics for this population.

Study design:

Observational study with minimal invasive procedures: population pharmacokinetic study.

Study population:

Critically ill children, admitted on the pediatric intensive care unit (PICU), receiving antibiotics.

Study parameters/endpoints:

Primary:

* To estimate population pharmacokinetic parameters for antibiotics

Secondary:

* To determine the target attainment rate of antibiotic exposure
* To design individualized dosing guidelines for antibiotics

Exploratory:

* To describe variability in kidney function
* To explore the relationship of genetic variation with disposition of pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 18 years of postnatal age;
* >37 weeks of gestational age (in children less than 6 months of postnatal age);
* Admitted to pediatric intensive care unit;
* Indwelling central line or arterial line in place for clinical purposes, or regular blood work for clinical reasons;
* Antibiotic therapy already prescribed by treating physician;
* Written informed consent (IC).

Exclusion Criteria:

* Language or cognitive inability to understand written and oral informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Critically ill children receiving antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Volume of distribution of antibiotics in critically ill children | 14 days
  Population mean value of volume of distribution of antibiotics during critical illness. Mean population volume of distribution will be derived from pooled data of antibiotic concentrations. Covariates of influence on volume of distribution will be incorporated within a population pharmacokinetic model.
Clearance of antibiotics in critically ill children | 14 days
  Population mean value of clearance of antibiotics during critical illness. Mean population clearance will be derived from pooled data of antibiotic concentrations. Covariates of influence on drug clearance will be incorporated within a population pharmacokinetic model.

CONTACTS AND LOCATIONS:
Overall Officials: Saskia N de Wildt, Prof. M.D., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hartman SJF, Upadhyay PJ, Mathot RAA, van der Flier M, Schreuder MF, Bruggemann RJ, Knibbe CA, de Wildt SN. Population pharmacokinetics of intravenous cefotaxime indicates that higher doses are required for critically ill children. J Antimicrob Chemother. 2022 May 29;77(6):1725-1732. doi: 10.1093/jac/dkac095. PMID 35383374
- [Derived] Hartman SJF, Upadhyay PJ, Hagedoorn NN, Mathot RAA, Moll HA, van der Flier M, Schreuder MF, Bruggemann RJ, Knibbe CA, de Wildt SN. Current Ceftriaxone Dose Recommendations are Adequate for Most Critically Ill Children: Results of a Population Pharmacokinetic Modeling and Simulation Study. Clin Pharmacokinet. 2021 Oct;60(10):1361-1372. doi: 10.1007/s40262-021-01035-9. Epub 2021 May 26. PMID 34036552